CLINICAL TRIAL: NCT05707585
Title: A Multicenter Study for Evaluating the Benign and Malignant Pulmonary Noldules by Detecting the Epigenetic Imprinting Alterations in Bronchoalveolar Lavage
Brief Title: Lung Cancer Diagnosis by Detecting Epigenetic Imprinting Alterations in Bronchoalveolar Lavage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Dalian Medical University (Other)
Collaborators: Fudan University (Other); Zongda Hospital affiliated to Southeast University (Network); West China Hospital (Other); Henan Provincial People's Hospital (Other); First Hospital of China Medical University (Other); Shengjing Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Lisen Imprinting Diagnostics, Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: LungCancerImprintingDiagnosis
Record Dates: First submitted 2023-01-19; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Lung Cancer
Keywords: Genomic Imprinting; Epigenetics; Diagnostic Study; Bronchoalveolar Lavage
MeSH Terms: conditions — Lung Neoplasms; Disease | interventions — In Situ Hybridization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Quantitative Chromogenic Imprinted Gene in situ Hybridization (QCIGISH) — Visualize and quantify the allelic expression status of imprinted genes by in situ hybridization using probes targeting the nascent RNAs

SUMMARY:
The goal of this multicenter observational study is to evaluate the lung cancer diagnostic value of epigenetic imprinting detection in bronchoalveolar lavage. This study will mainly focus on varifing the previously identified epigenetic imprinting biomarkers for lung cancer and upgrading and validating a lung cancer imprinting diagnostic model specifically for bronchoalveolar lavage. The lavage sample will be collected from each eligible paticipants under bronchialscopy and undergo QCIGISH detection to analyze the allelic expression status of imprinted genes. The QCIGISH detection results will be compared with the final surgical histopathology. No interventions will be taken according to the QCIGISH detection results.

DETAILED DESCRIPTION:
Bronchial biopsy and bursh are widely used in lung cancer diagnosis but not bronchoalveolar lavage because of its low sensitivity. As the molecular alterations usually occur before the morphological changes, genetic and epigenetic biomarkers will be helpful for early diagnosis of cancers. As an important epigenetic regulation in mammalian embryo development, genomic imprinting plays important roles in cancers. In normal post-natal somatic cells, imprinted genes are "silenced", that is mono-allelically expressed either from the maternal or paternal allele, while in cancers, some silenced imprinting genes' copies could be reactivated, leading to expressions from both alleles. The loss of monoallelic gene regulation is named loss of imprinting (LOI), and has been previously found in various human cancers. Our previous studies has identified several imprinted genes with elevated aberrant allelic expressions in lung cancer. A diagnostic model based on the epigenetic imprinting biomarkers achieved 99.1% sensitivity and 92.1% specificity. In this study, we will first verify the epigenetic imprinting biomarkers in bronchoalveolar lavage, and refine the previously developed diagnostic model specifically for lavage samples. The diagnostic model will be independently validated in a group of prospectively enrolled cases. This study will help to distinguish benign and malignant pulmonary nodules presurgically, and improve the early diagnosis of lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, and ≤ 75 years old;
* Chest CT showed pulmonary nodule with diameter<3cm;
* Subjects voluntarily participated and signed the informed consent form.

Exclusion Criteria:

* Active massive hemoptysis;
* Severe heart and lung dysfunction;
* Severe arrhythmia;
* Extreme exhaustion of general condition;
* Coagulation dysfunction;
* Acute attack of asthma;
* Aortic aneurysm.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary nodules and meet the criteria of bronchoscopy examination
Sampling Method: Probability Sample
Enrollment: 2064 (Estimated)
Dates: Start 2023-01-29 (Actual); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Epigenetic Imprinting Diagnostic Score | Within 10 days after each sample collected
  Cancer risk scores calculated by combining the biallelic expressions, multiallelic expressions and total expressions of several imprinted genes

CONTACTS AND LOCATIONS:
Overall Officials: Qi Wang, MD, Study Director — The Second Affiliated Hospital of Dalian Medical University
Locations (3):
- China (3):
  - Zongda Hospital affiliated to Southeast University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Zhongshan Hospital Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jelinic P, Shaw P. Loss of imprinting and cancer. J Pathol. 2007 Feb;211(3):261-8. doi: 10.1002/path.2116. PMID 17177177
- [Background] Bartolomei MS, Tilghman SM. Genomic imprinting in mammals. Annu Rev Genet. 1997;31:493-525. doi: 10.1146/annurev.genet.31.1.493. PMID 9442905
- [Background] Ribarska T, Goering W, Droop J, Bastian KM, Ingenwerth M, Schulz WA. Deregulation of an imprinted gene network in prostate cancer. Epigenetics. 2014 May;9(5):704-17. doi: 10.4161/epi.28006. Epub 2014 Feb 10. PMID 24513574
- [Background] Matouk IJ, Halle D, Gilon M, Hochberg A. The non-coding RNAs of the H19-IGF2 imprinted loci: a focus on biological roles and therapeutic potential in Lung Cancer. J Transl Med. 2015 Apr 9;13:113. doi: 10.1186/s12967-015-0467-3. PMID 25884481
- [Background] Ito Y, Koessler T, Ibrahim AE, Rai S, Vowler SL, Abu-Amero S, Silva AL, Maia AT, Huddleston JE, Uribe-Lewis S, Woodfine K, Jagodic M, Nativio R, Dunning A, Moore G, Klenova E, Bingham S, Pharoah PD, Brenton JD, Beck S, Sandhu MS, Murrell A. Somatically acquired hypomethylation of IGF2 in breast and colorectal cancer. Hum Mol Genet. 2008 Sep 1;17(17):2633-43. doi: 10.1093/hmg/ddn163. Epub 2008 Jun 9. PMID 18541649
- [Background] Shen R, Cheng T, Xu C, Yung RC, Bao J, Li X, Yu H, Lu S, Xu H, Wu H, Zhou J, Bu W, Wang X, Si H, Shi P, Zhao P, Liu Y, Deng Y, Zhu Y, Zeng S, Pineda JP, Lin C, Zhou N, Bai C. Novel visualized quantitative epigenetic imprinted gene biomarkers diagnose the malignancy of ten cancer types. Clin Epigenetics. 2020 May 24;12(1):71. doi: 10.1186/s13148-020-00861-1. PMID 32448196
- [Background] Xu H, Zhang Y, Wu H, Zhou N, Li X, Pineda JP, Zhu Y, Fu H, Ying M, Yang S, Bao J, Yang L, Zhang B, Guo L, Sun L, Lu F, Wang H, Huang Y, Zhu T, Wang X, Wei Q, Sheng C, Qu S, Lv Z, Xu D, Li Q, Dong Y, Qin J, Cheng T, Xing M. High Diagnostic Accuracy of Epigenetic Imprinting Biomarkers in Thyroid Nodules. J Clin Oncol. 2023 Feb 20;41(6):1296-1306. doi: 10.1200/JCO.22.00232. Epub 2022 Nov 15. PMID 36378996
- [Background] Zhou J, Cheng T, Li X, Hu J, Li E, Ding M, Shen R, Pineda JP, Li C, Lu S, Yu H, Sun J, Huang W, Wang X, Si H, Shi P, Liu J, Chang M, Dou M, Shi M, Chen X, Yung RC, Wang Q, Zhou N, Bai C. Epigenetic imprinting alterations as effective diagnostic biomarkers for early-stage lung cancer and small pulmonary nodules. Clin Epigenetics. 2021 Dec 14;13(1):220. doi: 10.1186/s13148-021-01203-5. PMID 34906185